CLINICAL TRIAL: NCT06169631
Title: The Effects of Noninvasive Brain Stimulation on Mental States, Behavior, and Electrophysiology
Brief Title: The Effects of Noninvasive Neuromodulation on Mental Wellness, Behavior, and Electrophysiology
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sanmai Technologies PBC dba Sanmai (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00064110
Record Dates: First submitted 2023-12-04; First posted 2023-12-13 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Anxiety Disorders
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Each experiment arm will have its own group(s).
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (3):
- Experiment 1 (Experimental): The study will consist of 2 groups. A: no current diagnosis of anxiety or other psychological disorders. B: Current diagnosis of anxiety disorder. Results will be analyzed within and between groups. Participants will answer standardized questionnaires and other similar validated psychological scales. An ultrasound transducer will be placed on their head aimed at the brain region of interest. EEG data will be collected throughout the process. After this process, participants will answer a set of post experiment questions.
  Interventions: Device: Gen0b
- Experiment 2a (Experimental): Current diagnosis of anxiety disorder is required. Participants will receive an MRI. Participants will answer standardized questionnaires and other similar validated psychological scales. An ultrasound transducer will be placed on their head aimed at the brain region of interest. EEG data will be collected throughout the process. After this process, participants will answer a set of post experiment questions
  Interventions: Device: Gen0b
- Experiment 2b (Experimental): Experiment 2b will expand on Experiment 2a protocol with multiple visits. Each visit will consist of the same activities as Experiment 2a.
  Interventions: Device: Gen0b

INTERVENTIONS:
Device: Gen0b — The ultrasound will be administered to the brain region of interest.

SUMMARY:
The purpose of the study is to test the effects of brief, low-intensity transcranial focused ultrasound (TUS) on electrophysiological, behavioral, and cognitive markers related to anxiety disorders.

DETAILED DESCRIPTION:
We will test the effects of TUS on self-reported and clinical anxiety states in healthy participants and in those with diagnosed anxiety disorders. Participants in these studies will receive pulsed TUS to the brain regions of interest. We will test whether multiple doses of TUS lead to larger reductions in mental states related to anxiety in comparison to a single dose of TUS.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years of age, as verified via photo identification with date of birth.
* Should be an English speaker, as indicated by being able to read and comprehend the consent form.
* Experiment 2 : Participants will be included for a past diagnosis of anxiety within the past year.

Exclusion Criteria:

* Smokes or uses tobacco products or any form of nicotine excessively
* History of head injury with loss of consciousness for more than 5 min
* Uncorrected hearing or vision impairment, including color blindness
* Currently have or history of brain or mental illness judged likely to interfere with testing, including drug and/or alcohol dependence
* History of epilepsy
* Brain tumors
* Takes medications or drugs judged likely to change brain activity, including psychoactive drugs, stimulants, benzodiazepines, and/or others
* Factors that may lead to poor EEG or fNIRS recordings (e.g., hairstyle)
* Inadequate sleep
* Drug, alcohol or prescription drug intoxication, dependence or addiction
* Pregnancy, or becoming pregnant during the course of the study
* Mild cognitive impairment or impaired decision making
* History of migraines
* Experience with neurostimulation (which might unbind or alter the results)
* Metal implants in their head or face

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-04-29 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Hamilton Anxiety Rating Inventory | 1 month
  Psychological questionnaire used by clinicians to rate the severity of a patient's anxiety

CONTACTS AND LOCATIONS:
Overall Officials: Jay Sanguinetti, PhD, Principal Investigator — Sanmai Technologies PBC; Taylor Kuhn, PhD, Principal Investigator — Sanmai Technologies PBC
Locations (1):
- Sanmai Technologies PBC, Sunnyvale, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tyler WJ. Noninvasive neuromodulation with ultrasound? A continuum mechanics hypothesis. Neuroscientist. 2011 Feb;17(1):25-36. doi: 10.1177/1073858409348066. Epub 2010 Jan 25. PMID 20103504
- [Result] Kubanek J. Neuromodulation with transcranial focused ultrasound. Neurosurg Focus. 2018 Feb;44(2):E14. doi: 10.3171/2017.11.FOCUS17621. PMID 29385924
- [Result] Fini M, Tyler WJ. Transcranial focused ultrasound: a new tool for non-invasive neuromodulation. Int Rev Psychiatry. 2017 Apr;29(2):168-177. doi: 10.1080/09540261.2017.1302924. Epub 2017 Apr 21. PMID 28430535
- [Result] Legon W, Bansal P, Tyshynsky R, Ai L, Mueller JK. Transcranial focused ultrasound neuromodulation of the human primary motor cortex. Sci Rep. 2018 Jul 3;8(1):10007. doi: 10.1038/s41598-018-28320-1. PMID 29968768
- [Result] Tufail Y, Matyushov A, Baldwin N, Tauchmann ML, Georges J, Yoshihiro A, Tillery SI, Tyler WJ. Transcranial pulsed ultrasound stimulates intact brain circuits. Neuron. 2010 Jun 10;66(5):681-94. doi: 10.1016/j.neuron.2010.05.008. PMID 20547127
- [Result] Sanguinetti JL, Hameroff S, Smith EE, Sato T, Daft CMW, Tyler WJ, Allen JJB. Transcranial Focused Ultrasound to the Right Prefrontal Cortex Improves Mood and Alters Functional Connectivity in Humans. Front Hum Neurosci. 2020 Feb 28;14:52. doi: 10.3389/fnhum.2020.00052. eCollection 2020. PMID 32184714
- [Result] Hameroff S, Trakas M, Duffield C, Annabi E, Gerace MB, Boyle P, Lucas A, Amos Q, Buadu A, Badal JJ. Transcranial ultrasound (TUS) effects on mental states: a pilot study. Brain Stimul. 2013 May;6(3):409-15. doi: 10.1016/j.brs.2012.05.002. Epub 2012 May 29. PMID 22664271
- [Result] Smith EE, Reznik SJ, Stewart JL, Allen JJ. Assessing and conceptualizing frontal EEG asymmetry: An updated primer on recording, processing, analyzing, and interpreting frontal alpha asymmetry. Int J Psychophysiol. 2017 Jan;111:98-114. doi: 10.1016/j.ijpsycho.2016.11.005. Epub 2016 Nov 17. PMID 27865882
- [Result] Kuhn T, Spivak NM, Dang BH, Becerra S, Halavi SE, Rotstein N, Rosenberg BM, Hiller S, Swenson A, Cvijanovic L, Dang N, Sun M, Kronemyer D, Berlow R, Revett MR, Suthana N, Monti MM, Bookheimer S. Transcranial focused ultrasound selectively increases perfusion and modulates functional connectivity of deep brain regions in humans. Front Neural Circuits. 2023 Apr 5;17:1120410. doi: 10.3389/fncir.2023.1120410. eCollection 2023. PMID 37091318